CLINICAL TRIAL: NCT05625659
Title: Comparison of Breast Cancer Screening With Dual-Energy Contrast-Enhanced Spectral Mammography to Digital Breast Tomosynthesis in Women With Dense Breasts (Contrast Mammography Imaging Screening Trial
Brief Title: Comparison of Breast Cancer Screening With CESM to DBT in Women With Dense Breasts
Acronym: CMIST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: American College of Radiology (Other)
Collaborators: GE Healthcare (Industry); Breast Cancer Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ACR A4707
Record Dates: First submitted 2022-11-15; First posted 2022-11-23 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: All participants who meet eligibility criteria will be offered Contrast Enhanced Spectral Mammography (CESM) in addition to their routine annual screening Digital Breast Tomosynthesis (DBT) at both the year 0 and year 1 visits.
Masking Description: Two independent readers at each institution participating in the trial will be assigned the task of either interpreting the results of the DBT images or the CESM images: one reader will read only the DBT images, while the other will read only the CESM images. Both individuals will be blinded to the results of the other modality, and the readers may not discuss their findings before both finalize their interpretations and complete the requisite CRFs.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DBT and CESM Diagnostic Imaging in Women with Dense Breasts (Other): Interventional Diagnostic
  Interventions: Diagnostic Test: Dual-Energy Contrast-Enhanced Spectral Mammography (CESM)

INTERVENTIONS:
Diagnostic Test: Dual-Energy Contrast-Enhanced Spectral Mammography (CESM) — In addition to their standard, digital breast tomosynthesis mammogram (DBT) performed at their regular screening visits, all participants will also receive a contrast-enhanced spectral mammography (CESM). These same diagnostic tests, both the DBT and CESM, with be repeated at 1 year post study entry for all participants. At year 2 post study entry, all participants will return to their usual breast screening exams and no longer received a CESM.

SUMMARY:
The over-arching goal of the Contrast-Enhanced Spectral Mammography Imaging Screening Trial (CMIST) is to determine if dual-energy contrast-enhanced spectral mammography (CESM) can detect more cancers with fewer false positives than digital breast tomosynthesis (DBT) in women with dense breasts.

Aim 1: To evaluate the performance of CESM compared to DBT at baseline for breast-cancer screening in women with dense breasts.

Aim 2: To evaluate the performance of CESM compared to DBT at the 1-year follow up for breast-cancer screening in women with dense breasts.

DETAILED DESCRIPTION:
The Contrast-Enhanced Spectral Mammography Imaging Screening Trial (CMIST), which will be managed by the American College of Radiology (ACR), Center for Research and Innovation (CRI), seeks to determine if dual-energy contrast-enhanced spectral mammography (CESM) screening provides more accurate cancer detection compared to digital breast tomosynthesis (DBT) in women with dense breasts.

Year 0 Visit:

All women aged 45 to 74 years of age known mammographically dense breasts, as reported on their most recent prior mammogram who are scheduled for a routine annual screening DBT will be offered CESM in addition to DBT. Baseline imaging (Year 0) will be performed within 30 days after participant registration. Standard DBT screening views followed by standard CESM screening views will be performed on the same day and prior to any additional workup.

Year 1 Visit (12 Months ±2 Months After Year 0 Imaging):

Standard DBT screening views followed by standard CESM screening views will be performed on the same day and prior to any additional workup.

Year 2 Visit: Follow-Up - Return for Standard Mammography Screening (12 Months ±2 Months After Year 1 Imaging):

The 2-year participant follow-up contact (email, text, or phone calls) should be performed 12 months (±2 months) after the Year 1 imaging to confirm the participant has not been diagnosed with an interval breast cancer. If 2-year imaging has not been scheduled, the 2-year participant follow-up contact should be performed prior to 14 months post year 1 visit. Participants diagnosed with breast cancer in the interval between the Year 1 and Year 2 imaging studies will have no subsequent follow-up and will not undergo the Year 2 study imaging in the scope of the study. The participant will be asked for AEs/SAEs with a non-leading question.

ELIGIBILITY:
Inclusion Criteria:

* 1. Women must have mammographically dense breasts, ACR BI-RADS® lexicon categories c or d (heterogeneous or extreme fibroglandular tissue) on their most recent prior screening.
* 2. Women agree to not undergo whole breast screening ultrasound for the duration of the trial until the year 2 standard of care imaging.
* 3. Women must not have symptoms or signs of benign or malignant breast disease (e.g., bloody, or clear nipple discharge, breast lump, focal breast pain).
* 4. Women must be able to undergo intravenous (IV) administration of iodinated contrast (e.g., no contraindication to intravenous contrast administration for Omnipaque [iohexol], and no known allergy-like reaction to iodine or moderate or severe allergic reactions to one or more allergens as defined by the American College of Radiology [ACR]: https://www.acr.org/-/media/ACR/files/clinical-resources/contrast_media.pdf).
* 5. Women must not be pregnant or breast-feeding. All females of childbearing potential who are uncertain if they could be pregnant or may be pregnant or as per local site standard of practice in women undergoing DBT and CESM must have a negative blood test or urine pregnancy test prior to Omnipaque (iohexol) administration. A female of childbearing potential is any woman, regardless of sexual orientation, sexual identity or whether they have undergone tubal ligation, who meets the following criteria: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months).
* 6. Women of childbearing potential must be strongly advised to use an accepted and effective method of contraception or to abstain from sexual intercourse for the following year until the Year 1 DBT and CESM studies are performed.

Exclusion Criteria:

* 1. Women currently undergoing treatment for breast cancer, or planning surgery for a high-risk lesion (ADH, ALH, LCIS, papilloma, radial scar).
* 2. Women who have had the following are not eligible:

  1. a mammogram less than 11 months prior to study entry.
  2. screening breast ultrasound within 11 months prior to study entry.
  3. breast MRI less than 36 months prior to study entry.
  4. contrast-enhanced spectral mammography less than 36 months prior to study entry.
  5. molecular breast imaging (MBI) less than 36 months prior to study entry.
  6. breast prosthetic implants (silicone or saline).
  7. suspected of being at high-risk for breast cancer, as defined by the ACS breast MR screening recommendations (lifetime risk of ≥20%-25%) unless they are unable to undergo an MRI. (Reference Appendix I)
  8. a history of sickle cell disease.
* 3. Women with known or suspected renal impairment. Requirements for glomerular filtration rate (GFR) determination prior to IV iodinated contrast administration are determined by local site standard practice. Criteria that should be considered include, but are not limited to, the following:
* Age >60 years old
* History of renal disease, including dialysis, kidney transplant, single kidney, renal cancer, and renal surgery
* History of hypertension requiring medical therapy
* History of diabetes mellitus
* Use of metformin or metformin-containing drug combinations
* 4. Women who are pregnant, breast feeding, or planning to become pregnant from screening until 30 days after the last administration of Omnipaque (iohexol).
* 5. Large breasted women that require multiple images per standard view of the breast (Tiling) as determined by their most recent mammogram.

Ages: 45 Years to 74 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2032 (Estimated)
Dates: Start 2023-03-24 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Cancer Detection Rate | Year 0
  The cancer detection rate (CDR) at the participant level at Year 0. This measure will be evaluated for CESM and DBT
Recall Rate | 1 Year
  The recall rate for participants at Year 1, which will be estimated for each imaging modality separately.

CONTACTS AND LOCATIONS:
Locations (10):
- United States (9):
  - University of Alabama, Birmingham, Birmingham, Alabama
  - Boca Raton Regional Hospital - Christine E. Lynn Women's Health and Wellness Institute, Boca Raton, Florida
  - Lake Medical Imaging, The Villages, Florida
  - Henry Ford Health, Detroit, Michigan
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Carolina Breast Imaging Specialists, Greenville, North Carolina
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - University of Virginia, Charlottesville, Virginia
- St. Joseph's Hospital, London, Ontario, Canada